CLINICAL TRIAL: NCT03159767
Title: Validation of a New Method of Measuring Spinal Flexibility in Axial Spondyloarthritis Using Inertial Motion (IMU) Sensors
Brief Title: A Clinimetric Test of Spinal Sensors in Measuring Spinal Mobility in Axial Spondyloarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Philip Gardiner (Other)
Collaborators: University of Ulster (Other)
Responsible Party: Sponsor-Investigator, Dr Philip Gardiner, Consultant Rheumatologist, Western Health and Social Care Trust
Organization: Western Health and Social Care Trust (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: WT 15/28
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Ankylosing Spondylitis; Axial Spondyloarthritis
MeSH Terms: conditions — Spondylitis, Ankylosing; Axial Spondyloarthritis

STUDY DESIGN:
Intervention Model Description: Clinimetric study comparing repeated standardised spinal mobility test protocols by two independent raters on two occasions
Who Masked: Outcomes Assessor
Masking Description: Each physiotherapist rater will have to independently attach the sensors to the participant's spine before testing, and no positioning marks will be left on the patient in between tests or between visits. They will work in different rooms and will not have access to earlier results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal Mobility Measurement: Rater A (Experimental): All patients will undergo the same ViMove Spinal Sensor measurement protocol with independent raters.
  Interventions: Device: ViMove Spinal Sensor
- Spinal Mobility Measurement: Rater B (Experimental): All patients will undergo the same ViMove Spinal Sensor measurement protocol with independent raters.
  Interventions: Device: ViMove Spinal Sensor

INTERVENTIONS:
Device: ViMove Spinal Sensor — Sensors will be used to measure spinal movement

SUMMARY:
This is a clinimetric study to validate the use of IMU spinal sensors to measure the range of spinal movement in a group of patients with axial spondyloarthritis.

DETAILED DESCRIPTION:
One of the most important goals of therapy in axial spondyloarthritis is to improve and/or preserve spinal mobility. In the early stages of the disease, spinal stiffness is reversible but eventually the spine can fuse causing permanent loss of flexion. Traditional tests for spinal mobility using tape measures are inaccurate and do not capture many aspects of kinematics such as spinal rotation or speed of movement. There is also a need for wearable sensors to give patients feedback and encourage more regular exercise.

The investigators will be using IMU spinal sensors to measure spinal ROM in a group of 40 patients with axial spondyloarthritis. The investigators will be testing aspects of inter-rater and intra-rater reliability, comparing sensor reliability to the accuracy of the traditional tape measure test (BASMI).

ELIGIBILITY:
Inclusion Criteria:

-Confirmed diagnosis of axSpA according to the ASAS criteria

Exclusion Criteria:

* Severe joint or spinal pain at the time of the study
* Severely restricted hip movement
* History of previous vertebral fracture
* History of previous spinal surgery
* Major scoliosis deformity
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Inter-rater reliability for measurement of lumbar spine range of movement | 2 weeks
  ICC for lumbar side flexion and forward flexion expected to be >0.8

SECONDARY OUTCOMES:
Inter-rater reliability for measurement of lumbar spine rotational range of movement | 2 weeks
  ICC for spinal rotation expected to be >0.8
Reliability of IMU metrology index non-inferior to reliability of BASMI | 2 weeks
  Measurements obtained using IMUs are at least as reliable as the BASMI tape measure test
Correlation with BASDAI: IMU metrology index non-inferior compared to BASMI | 2 weeks
  We will compare the metrology indices in the strength of correlation with the BASDAI components of pain and stiffness.
Inter-rater reliability for measurement of cervical rotation range of movement | 2 weeks
  ICC for cervical rotation expected to be >0.8

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gardiner, MD, Principal Investigator — Western HSCT
Locations (1):
- Department of Rheumatology, Altnagelvin Hospital, Londonderry, N.Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: No